CLINICAL TRIAL: NCT06801262
Title: TreaT-Assay: the New Frontier for the Diagnosis of Acute Rejection in Kidney Transplantation
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TreaT2021
Record Dates: First submitted 2024-12-30; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Kidney Diseases; Kidney Transplant; Kidney Disease, End-Stage
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Basic hematochemical evaluation. These examinations belong to the type of tests normally performed for biochemical and laboratory follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kidney transplantation is the standard therapy for end-stage renal disease. Acute rejection (AR) or chronic rejection along with reactive donor immunity, which counteracts organ acceptance, are among the greatest medical challenges in transplantation.

In the posttransplantation setting, immunosuppressive drugs are administered to control or prevent immune reactions; however, the therapies have serious side effects. Retrospective studies have shown heterogeneous risk profiles with respect to post-transplant complications, such as AR or infection, suggesting the introduction of an individualized immunosuppressive regimen2,3,4. Biomarkers are needed for such individual therapies to discriminate between patients with different risk profiles.

DETAILED DESCRIPTION:
Kidney transplantation is the standard therapy for end-stage renal disease. Acute rejection (AR) or chronic rejection along with reactive donor immunity, which counteracts organ acceptance, are among the greatest medical challenges in transplantation.

In the posttransplantation setting, immunosuppressive drugs are administered to control or prevent immune reactions; however, the therapies have serious side effects. Retrospective studies have shown heterogeneous risk profiles with respect to post-transplant complications, such as AR or infection, suggesting the introduction of an individualized immunosuppressive regimen. Biomarkers are needed for such individual therapies to discriminate between patients with different risk profiles.

The presence of donor reactive T-cells pre and post kidney transplantation correlates with acute rejection and with reduced allograft survival1,7,8. For these reasons, a specific and sensitive assay has been developed for in-depth monitoring and characterization of reactive T cells from allografts: the Transplant reactive T-cells-assay (TreaT assay). For the latter, donor TECs, obtained from the recipient's urine by selective catherization of the transplanted kidney, a useful and renewable antigenic source for stimulation of recipient PBMCs, are used as the stimulating source.

The TreaT assay, compared with previous tests, has the advantages of unlimited availability of starting sample, easy in implementation, inexpensive and superior performance. Pilot studies, have obtained encouraging data on the test's applicability in patients with early acute rejection and prediction of post-transplant eGFR. In addition, this approach provides insight into the biology of alloreactive immune cells specifically, the immunological interaction with donor/recipient in post-transplantation. Therefore, it could help guide a personalized pharmacological approach of therapy in the future of kidney transplantation.

The study is non-interventional and requires obtaining clinical data from recruited subjects and blood and urine samples. Therefore, no added risk to the subjects involved is expected.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for subjects in group A Healthy adult subjects who will be selected from blood donors belonging to the Metropolitan Immunohematology and Transfusion Medicine Service. It should be noted that for subjects belonging to group A, informed consent is not required as the samples are provided in anonymous manner and completely unrelated to the patient.
* Inclusion criteria for study patients group B

  1. Subjects undergoing living or cadaveric kidney transplantation afferent to the O.U. of Nephrology, Dialysis and Renal Transplantation, St. Orsola Hospital, Pavilion 15.
  2. Patients who intend to participate in the study.

Exclusion Criteria:

* Exclusion criteria for subjects in group A None
* Exclusion criteria for patients in study group B

  1. Subjects under the age of 18 years.
  2. Patients who are unable to make explicit their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing living and cadaveric kidney transplantation will be considered, afferent to the Department of Nephrology at St. Orsola Hospital, Pavilion 15, who meet the criteria of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Create the TreaT test | 5 years
  The study aims to create a pivotal tool (the TreaT test) by collecting and culturing PBMCs and TECs from kidney transplant recipient.

SECONDARY OUTCOMES:
Identification of reactive T cells involved in acute rejection | T0 (pre-transplant), T1 (first week post-transplant), T2(3 months) and T3 (6 months)
  Assess the various lymphocyte subpopulations: Th1, Th2, Th17, natural killer, Treg, Memory, monocytes and B cells and the production of pro- and anti-inflammatory cytokines following co-culture with TEC
Understand the immunological and molecular basis of acute rejection and predictive markers | T0 (pre-transplant), T1 (first week post-transplant), T2(3 months) and T3 (6 months)
  Biomarkers, via TreaT assay, with high positive and/or negative predictive value, sensitive and minimally invasive will be sought. The strategy, termed "unbiased," implemented for the identification of new biomarkers, is the screening of proteins, genes, etc. not based on any specific hypothesis except that through these assays it will be possible to identify elements capable of differentiating groups of subjects with distinct clinical phenotypes.
Search for markers for acute rejection | T0 (pre-transplant), T1 (first week post-transplant), T2(3 months) and T3 (6 months)
  Evaluation of the correlation of potential instrumental, laboratory markers (lymphocyte subpopulations, plasma, serum and urinary concentrations of previously identified predictive markers) with the presence and type of histologically demonstrated acute rejection and specific histologic lesions (according to Banff 2017 classification).

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano La Manna, MD, Principal Investigator — IRCCS Azienza Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy